CLINICAL TRIAL: NCT05931250
Title: Alternating and Direct Current Stimulation for the Treatment of Chronic Neuropathic Eye Pain and Cerebral Symptoms: a Pilot Study
Brief Title: Alternating and Direct Current Stimulation for Neuropathic Eye Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neil Lagali (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor-Investigator, Neil Lagali, Principal Investigator, Professor, Region Östergötland
Organization: Region Östergötland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220727401
Record Dates: First submitted 2023-06-16; First posted 2023-07-05 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Eye Pain; Neuropathy, Optic; Cerebral Injury
MeSH Terms: conditions — Eye Pain; Optic Nerve Diseases; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial alternating current stimulation (Experimental): Transcranial alternating current stimulation (tACS) device using 50x70 mm electrodes that are placed bilaterally between EEG coordinates C3/C5 for left hemisphere and C4/C6 for right hemisphere (corresponding to S1 and M1 of the eye). The alternating current electrodes are in-phase and have the same peak to peak stimulation 3mA, for 30 minutes duration at 10Hz. An impedance value under 15 ohms is required at all times to ensure patient comfort and safety.
  Interventions: Device: DC-Stimulator Plus (NeuroConn GmbH, Germany)
- Transcranial direct current stimulation (Experimental): Transcranial direct current stimulation (tDCS) device using 50x70 mm electrodes that has the anodal electrode placed contralateral to most prominent ocular pain or, in the case of bilateral pain symptoms, contralateral to the dominant hand between EEG coordinates C3/C5 for left hemisphere and C4/C6 for right hemisphere (corresponding to S1 and M1 of the eye), and the cathode placed on the patient's upper arm. A current peaking at 3mA will ramp up for 20 secs and be delivered for a total of 20 minutes, thereafter, ramping down for 20s. An impedance value under 15 ohms is required at all times to ensure patient comfort and safety.
  Interventions: Device: Sooma direct current stimulator (Sooma, Finland)

INTERVENTIONS:
Device: DC-Stimulator Plus (NeuroConn GmbH, Germany) — Transcranial alternating current stimulation
  Arms: Transcranial alternating current stimulation
Device: Sooma direct current stimulator (Sooma, Finland) — Transcranial direct current stimulation
  Arms: Transcranial direct current stimulation

SUMMARY:
The goal of this clinical intervention is to test if two forms of transcranial current stimulation, transcranial direct current stimulation (tDCS) or transcranial alternating current stimulation (tACS) can alleviate neuropathic eye pain in a sample of 20 patients.

The main aims are:

* Test if tDCS/tACS can alleviate neuropathic eye pain and/or other cerebral symptoms: brain fatigue, migraine, light sensitivity, etc.
* Test if one stimulation method is superior to the other Patients will be treated for a total of fifteen 30-minute stimulation sessions, three times a day over a five-day period, each stimulation separated by approximately 4 hours, with either active tACS or tDCS over the scalp corresponding to primary sensory and motor areas.

The patients will have questionnaires to monitor subjective experiences and pupillometry before and after treatment to monitor experimental outcomes.

DETAILED DESCRIPTION:
Brief Summary sufficient

ELIGIBILITY:
Inclusion Criteria:

* persistent eye pain for at least 6 months
* average eye pain intensity of 4 or more on a 0-10 numerical rating scale
* naive to transcranial stimulation
* eye pain having neuropathic-like characteristics

Exclusion Criteria:

* contraindication to transcranial stimulation (i.e., pacemaker, cardioverter defibrillator, neuro-stimulation (brain or spinal cord), bone growth stimulations, indwelling blood pressure monitors, epilepsy, pregnancy)
* presence of ocular diseases that are the likely cause of pain (i.e., corneal and conjunctival scarring, corneal edema, uveitis, iris transillumination defects, etc.)
* current participation in another study with an investigational drug or device within one month prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline subjective pain via neuropathic pain symptom inventory for the eye (NPSI-eye) at 1 week | through treatment completion, 1 week
  Assesses pain related symptoms on a scale from 0 indicating no pain (better outcome) to10 indicating worst pain imaginable (worse outcome)
Change from baseline subjective pain via neuropathic pain symptom inventory for the eye (NPSI-eye) at 2 weeks | through treatment completion, 2 weeks
  Assesses pain related symptoms on a scale from 0 indicating no pain (better outcome) to10 indicating worst pain imaginable (worse outcome)
Change from baseline subjective pain via neuropathic pain symptom inventory for the eye (NPSI-eye) at 1 month | through treatment completion, 1 month
  Assesses pain related symptoms on a scale from 0 indicating no pain (better outcome) to10 indicating worst pain imaginable (worse outcome)
Change from baseline subjective pain effect experiences via Defense and Veteran Pain Rating Scale (DVPRS) at 1 week | through treatment completion, 1 week
  Assesses pain related symptoms effecting sleep, stress, disposition, life quality, on a scale from 0 indicating no effect (better outcome) to10 indicating maximum effect (worse outcome)
Change from baseline subjective pain effect experiences via Defense and Veteran Pain Rating Scale (DVPRS) at 2 weeks | through treatment completion, 2 weeks
  Assesses pain related symptoms effecting sleep, stress, disposition, life quality, on a scale from 0 indicating no effect (better outcome) to10 indicating maximum effect (worse outcome)
Change from baseline subjective pain effect experiences via Defense and Veteran Pain Rating Scale (DVPRS) at 1 month | through treatment completion, 1 month
  Assesses pain related symptoms effecting sleep, stress, disposition, life quality, on a scale from 0 indicating no effect (better outcome) to10 indicating maximum effect (worse outcome)
Change from baseline subjective mental symptoms via Mental Fatigue Scale (MFS) at 1 week | through treatment completion, 1 week
  Assesses mental symptoms on a scale from 0 indicating no effect (better outcome) to 3 indicating extreme effect (worse outcome)
Change from baseline subjective mental symptoms via Mental Fatigue Scale (MFS) at 2 weeks | through treatment completion, 2 weeks
  Assesses mental symptoms on a scale from 0 indicating no effect (better outcome) to 3 indicating extreme effect (worse outcome)
Change from baseline subjective mental symptoms via Mental Fatigue Scale (MFS) at 1 month | through treatment completion, 1 month
  Assesses mental symptoms on a scale from 0 indicating no effect (better outcome) to 3 indicating extreme effect (worse outcome)
Change from baseline subjective ocular symptoms and symptom frequency via custom ocular pain questionnaire at 1 week | through treatment completion, 1 week
  Ocular pain questionnaire using a visual analog scale with 0 indicating no pain (better outcome) and 10 indicating extreme pain (worse outcome) and frequency measure from 0% indicating never occurring (better outcome) to 100% indicating always occurring (worse outcome)
Change from baseline subjective ocular symptoms and symptom frequency via custom ocular pain questionnaire at 2 weeks | through treatment completion, 1 month
  Ocular pain questionnaire using a visual analog scale with 0 indicating no pain (better outcome) and 10 indicating extreme pain (worse outcome) and frequency measure from 0% indicating never occurring (better outcome) to 100% indicating always occurring (worse outcome)
Change from baseline subjective ocular symptoms and symptom frequency via custom ocular pain questionnaire at 1 month | through treatment completion, 1 month
  Ocular pain questionnaire using a visual analog scale with 0 indicating no pain (better outcome) and 10 indicating extreme pain (worse outcome) and frequency measure from 0% indicating never occurring (better outcome) to 100% indicating always occurring (worse outcome)
Number of patients with treatment-related adverse events as assessed by ocular pain questionnaire | through treatment completion, 1 month
  Ocular pain questionnaire using a visual analog scale with 0 indicating no pain (better outcome) and 10 indicating extreme pain (worse outcome) and frequency measure from 0% indicating never occurring (better outcome) to 100% indicating always occurring (worse outcome)
Change from baseline pupil diameter in millimeters at 1 week | through treament completion, 1 week
  Minimum and maximum pupil diameter in millimeters
Change from baseline pupil velocity in millimeters per second at 1 week | through treament completion, 1 week
  Pupil change velocity in millimeters per second
Change from baseline pupil latency in milliseconds at 1 week | through treament completion, 1 week
  Pupil latency latency in milliseconds

SECONDARY OUTCOMES:
Treatment compliance rate | through study completion, 1 year
  Evaluation of completed treatment from a total of 15

OTHER OUTCOMES:
Beta coefficients for participant demographics (sex, age, race/ethnicity) in regression model predicting adherence to treatment protocol | through study completion, 1 year
  Exploratory regression analysis to identify associations between demographic variables and number of treatment sessions completed
Beta coefficients for participant demographics (sex, age, race/ethnicity) in regression model predicting change in pain (Numerical Rating Scale) | through study completion, 1 year
  Exploratory regression analysis to identify associations between demographic variables and change in pain ratings (before vs. after stimulation treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Lagali, PhD, Principal Investigator — RegionÖstergötland
Locations (1):
- Eye Clinic, University Hospital in Linköping, Linköping, Other / Non-US, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qazi Y, Hurwitz S, Khan S, Jurkunas UV, Dana R, Hamrah P. Validity and Reliability of a Novel Ocular Pain Assessment Survey (OPAS) in Quantifying and Monitoring Corneal and Ocular Surface Pain. Ophthalmology. 2016 Jul;123(7):1458-68. doi: 10.1016/j.ophtha.2016.03.006. Epub 2016 Apr 16. PMID 27089999
- [Background] Farhangi M, Feuer W, Galor A, Bouhassira D, Levitt RC, Sarantopoulos CD, Felix ER. Modification of the Neuropathic Pain Symptom Inventory for use in eye pain (NPSI-Eye). Pain. 2019 Jul;160(7):1541-1550. doi: 10.1097/j.pain.0000000000001552. PMID 30883524
- [Background] Sivanesan E, Levitt RC, Sarantopoulos CD, Patin D, Galor A. Noninvasive Electrical Stimulation for the Treatment of Chronic Ocular Pain and Photophobia. Neuromodulation. 2018 Dec;21(8):727-734. doi: 10.1111/ner.12742. Epub 2017 Dec 28. PMID 29283468